CLINICAL TRIAL: NCT03418285
Title: Microbiota-derived Trimethylamine N-oxide as Residual Risk After ST-elevation Myocardial Infarction
Brief Title: Trimethylamine N-oxide in Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Yokohama City University Medical Center (Other)
Responsible Party: Principal Investigator, Yasushi Matsuzawa, MD. PhD., Yokohama City University Medical Center
Other Study IDs: TMAO_STEMI
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Trimethylamine-N-oxide (TMAO) is produced from the metabolism of gut microbiota and is reportedly pro-atherogenic and associated with cardiovascular events. The purpose of this study is to investigate the sequential change in TMAO levels by current optimal secondary prevention therapies in patients with ST-elevation acute myocardial infarction (STEMI) and the clinical impact of TMAO levels on the progression of atherosclerosis and subsequent cardiovascular events.

DETAILED DESCRIPTION:
This study includes patients with their first STEMI. The investigators measure plasma TMAO levels using the frozen plasma at the onset of STEMI and 10 months later (the chronic phase). To assess plaque progression, residual SYNTAX (Synergy Between Percutaneous Coronary Intervention With Taxus and Cardiac Surgery) score and chronic-phase SYNTAX score are measured. After the chronic-phase assessment of TMAO and SYNTAX score, patients are followed for cardiovascular events including death, myocardial infarction, ischemic stroke, and unstable angina pectoris with coronary revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Patients who admitted to the Yokohama City University Medical Center with the diagnosis of their first STEMI and who underwent primary percutaneous coronary intervention within 12 hours after onset and received follow-up coronary angiogram 10 months after the index intervention.

Exclusion Criteria:

* none

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
MACE | 6 years
  death, myocardial infarction, ischemic stroke, and unstable angina pectoris with coronary revascularization

SECONDARY OUTCOMES:
Coronary plaque progression | 10 months
  the highest tertile of change in SYNTAX (Synergy Between Percutaneous Coronary Intervention With Taxus and Cardiac Surgery) score.
  Higher SYNTAX score indicates more complicated coronary plaque. minimum 0, maximum 80.

IPD SHARING:
Plan to Share IPD: No